CLINICAL TRIAL: NCT05823038
Title: Evaluation of Implant Patients by Peri-implant Disease Risk Analysis and Aesthetic Score
Brief Title: Risk and Aesthetic Assesment in Implant Patient
Acronym: EIPPDRAAS
Status: Completed | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Tuğba ŞAHİN, Assistant professor, Abant Izzet Baysal University
Other Study IDs: 2022/160
Record Dates: First submitted 2023-04-08; First posted 2023-04-21 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-02

CONDITIONS: Implant Assesment
Keywords: Implant disease risk assesment; Pink esthetic score; Implant quality scale; Periodontal health; Periodontal disease
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study examines the peri-implant risk assessment diagram and the aesthetic, peri-implant health status, and gingival level around the implant in patients with implants by comparing them in smokers and non-smokers.

: After completion of the examination, 298 dental implants for at least three months after functional prosthesis loading, except for patients with bruxism and uncontrolled diabetes, were included in the study. Patients are primarily divided into smokers and non-smokers. In all implant patients, plaque, gingival index, bleeding on probing, pocket depth, clinical attachment loss, gingival recession, keratinized thickness, keratinized width, vestibule depth, pink aesthetic score, and peri-implant disease risk analysis are evaluated in sequence.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old patients
* Patients who are systemically healthy and have a controlled medical condition
* Patients with fixed prosthesis on the implant at least 6 months after the functional prosthetic loading of the dental implant

Exclusion Criteria:

* Patients with uncontrolled systemic diseases
* Those who have the habit of bruxism

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 298 dental implants for at least 6 months after functional prosthetic loading were included in the study. Patients are primarily divided into smokers and non-smokers.
Sampling Method: Probability Sample
Enrollment: 298 (Actual)
Dates: Start 2022-07-04 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-01-05 (Actual)

PRIMARY OUTCOMES:
Implant disease risk assesment | baseline
  The IDRA algorithm is a promising tool to assess patients at moderate or high risk of developing peri-implantitis. The eight vectors of the diagram include: an assessment of a history of periodontitis, the percentage of sites with bleeding on probing (BOP), the number of teeth/implants with probing depths (PD) ≥5 mm, the ratio of periodontal bone loss (evaluated from a radiograph) divided by the patient's age, periodontitis susceptibility as described by the staging and grading categories from the 2017 World Workshop on the Classification of Periodontal and Peri-implant Diseases , the frequency/compliance with supportive periodontal therapy, the distance from the restorative margin of the implant-supported prosthesis to the marginal bone crest, and prosthesis related factors including cleanability and fit of the implant-supported prosthesis.
Pink esthetic scale | baseline
  With the pink aesthetic score, the post-implant process is scored according to the papilla, tissue contours, gingival level, alveolar process, color, and tissue condition. The thresholds for clinical acceptance, which was currently set at values of 8/14 for the PES. The thresholds for clinical acceptance are currently set at values of 8 to 14 for the PES.
Dental implant health scale | baseline
  The Implant Quality of The Health Scale allows the dentist to evaluate an implant using the listed criteria, place it in the appropriate category of health or disease, and then treat the implant accordingly. Three primary classes were established by the Consensus: success, survival, and failure. The success category describes optimum conditions, the survival category describes implants still in function but not with ideal conditions, and the loss of an implant represents an the implant that should be or already has been removed.
  Implant Quality Scale Group Clinical Conditions
  1. Success (optimum health) a) No pain or tenderness upon function b) 0 mobility c) <2 mm radiographic bone loss from initial surgery d) No exudates history
  2. Satisfactory survival a) No pain on function b) 0 mobility c) 2-4 mm radiographic bone loss d) No exudates history
  3. Compromised survival a) May have sensitivity on function b) No mobility c) Radiographic bone loss> 4 mm(less than ½ of implant
Keratinized tissue thickness | baseline
  It is advanced to the bone with a canal file. The distance between the stopper and the tip of the file is measured.
Keratinized tissue width | baseline
  Keratinized mucosa width was defined as the distance between the gingival margin and mucogingival junction at the mid-buccal area
Periodontal depth | baseline
  Measuring the distance from the gingival margin to the mucogingival line with a periodontal probe.
Bleeding on probing | baseline
  To determine the bleeding index on probing, the pocket floor, and the inflammatory state of the pocket epithelium, an evaluation is made according to whether there is bleeding in the sulcus 30 seconds after the pocket depth measurement from 6 regions of all the teeth of the patients: mesiobuccal, mid-buccal, distobuccal, mesiolingual, mid-lingual and distolingual.
Vestibular depth | baseline
  Vestibular depth is measured either from crest of lip or from coronal border of the attached gingiva to depth of mucobuccal fold.

SECONDARY OUTCOMES:
Plaque index | baseline
  In the plaque index, the mesiobuccal, mid-buccal, distobuccal, mesiolingual, mid-lingual, and distolingual regions of the implant or implants and dental plaque thickness to the gingiva are evaluated by probing.
Gingival index | baseline
  The gingival index evaluates bleeding, the most basic sign of inflammation. The implants' mesiobuccal, mid-buccal, distobuccal, mesiolingual, mid-lingual, and distolingual surfaces are measured.
Clinical attachment level | baseline
  Clinical attachment level/loss measured in mm as distance from the CEJ to the gingival margin.
Gingival recession | baseline
  Gingival recession is the exposure of the root surface resulting from migration of the gingival margin apical to the cementoenamel junction.

CONTACTS AND LOCATIONS:
Overall Officials: Ramazan Kurul, Ass. Prof, Principal Investigator — Abant Izzet Baysal University
Locations (1):
- Bolu Abant İzzet Baysal University, Bolu, Turkey, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided